CLINICAL TRIAL: NCT00609713
Title: Bone Health of Obese Adolescents During Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-10-4976; 1R01HD049701-01A2 (NIH)
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Pediatric Obesity
Keywords: Child; Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Comprehensive 12-month family-based obesity treatment with separate adolescents and parents group sessions
  Interventions: Behavioral: Comprehensive behavioral weight control program
- 2 (Active Comparator): Individual 12-month nutrition education program
  Interventions: Other: Individual 12-month nutrition education program

INTERVENTIONS:
Behavioral: Comprehensive behavioral weight control program — Participants will meet weekly for 12 weeks, then every other week for 12 weeks, and once a month thereafter through week 52. Adolescents and parents will receive manuals that provide lessons and homework assignments for each meeting. The program for the first 22 weeks includes the following topics: 1) the causes of obesity; 2) components of healthy nutrition; 3) self-monitoring of calories, physical activity, and inactivity; 4) stimulus control procedures; 5) coping with high-risk social or psychological situations that trigger excess eating; 6) increasing physical activity; and 7) minimizing inactivity. At each session, participants will submit their self-monitoring diaries and completed homework. Incentives for completion of self-monitoring tasks are an integral part of the behavior modification program and a small gift certificate will be given to subjects for successful completion at each intervention session.
  Arms: 1
Other: Individual 12-month nutrition education program — The other half of the participants (44 subjects) will be randomized to this arm of the intervention (usual care), which will also start in five waves. In contrast to the comprehensive behavioral weight control program, the nutrition education program will take place through individual appointments with a clinical dietician to reflect usual care and mimic the present approach used for the treatment of obese adolescents at the Children's Hospital of Philadelphia (CHOP) Nutrition Consultation. Parents will be required to take part in the consultations. The first consultation will last 60 minutes and the following consultations of 30 minutes will take place once a month for the first six months, then every other month for the second six months, as is the usual practice in our clinical setting.
  Arms: 2

SUMMARY:
The long-term goal of this proposal is to understand the impact of obesity and obesity treatment on bone health during adolescence and how to preserve it. The recent pediatric obesity epidemic raises important clinical and public health questions about the effects of childhood-onset obesity and its treatment on bone health. Osteoporotic fractures are a major cause of morbidity and mortality in the aged, and peak bone mass (PBM), achieved shortly after puberty, is a key determinant of bone strength and lifetime fracture risk. Given the current obesity epidemic, obesity treatment during adolescence will continue to be necessary. The benefits of pediatric obesity treatment are unquestionable. However, the potential detrimental effects of weight loss on bone density and dimensions are not known in adolescents and are the focus of this proposal.

This study will focus on the impact of pediatric-onset obesity and its treatment on bone health, using two approaches: comparing obese and non-obese adolescents and comparing obese adolescents before and after weight loss. We hypothesize that (a) compared to non-obese controls, obese adolescents have stronger bones, and that (b) bone strength of obese adolescents decreases during weight loss compared to usual care, which would suggest a need to promote bone health during successful weight loss in obese adolescents.

DETAILED DESCRIPTION:
Context: The childhood obesity epidemic raises important clinical and public health questions about the effects of both obesity and obesity treatment on bone development. Osteoporotic fractures are a major cause of morbidity and mortality in the aged. However, peak bone mass, achieved shortly after puberty, is the key determinant of lifetime osteoporotic fracture risks. The size and direction of effects of obesity and weight loss on bone health in childhood are unclear, partly because of bone ascertainment issues. Obese children and adolescents may have elevated fracture risks, contrary to expectations based on adult data. Objectives: Primary aims of the proposed study are to: 1) characterize and compare bone health of obese and non-obese adolescents using the most accurate methods available, and 2) investigate the impact of comprehensive behavior weight control program on the bone health of obese adolescents. Study Design: Aim 1 will use a case-control design to compare bone status measures of 88 obese adolescents (ages 10 to 14 years), to be recruited for a randomized obesity treatment trial, with the same measurements of 51 contemporary non-obese control adolescents. For Aim 2, the 88 obese adolescents will be enrolled in a 12-month randomized trial, with 1:1 assignment, of a comprehensive behavioral weight control program vs. individualized nutrition education (usual care). This randomized trial is the object of this registration. Study Measures: For both aims the primary outcome will be bone strength, estimated by stress-strength index, and measured by peripheral quantitative computerized tomography (pQCT) at the tibia, a weight-bearing site.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be 10.0 to 14.9 years of age, with a body mass index (BMI) above the 97th percentile for age (~ +1.88 SD) and below +3.00 SD or less than 300 lb (~ 136 kg), whichever is lower.

Exclusion Criteria:

1. Syndromic or secondary obesity,
2. Developmental delay requiring special education,
3. Depression, psychosis,
4. Eating disorders that involve insufficient or excessive food intake, such as anorexia nervosa or bulimia,
5. Orthopedic problems interfering with moderate to vigorous physical activity,
6. Diabetes,
7. Polycystic ovary syndrome,
8. History of systemic corticosteroids use for more than three months cumulatively, use of immunomodulators, anticonvulsivants, weight loss medications (including diet supplements) and any other medications, or chronic conditions that could interfere with the intervention or with bone health.
9. Weight loss in the preceding six months of 5% or more, participation in another weight loss program,
10. Cigarette smoking (smoking and smoking cessation can affect weight and bones),
11. Sexual activity without contraception and/or pregnancy,
12. Subjects without a primary care provider or with a provider unwilling to provide to the research team medical information on the child will be excluded.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2007-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Quantitative computerized tomography (pQCT) | Base line, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Babette Zemel, PhD, Principal Investigator — CHOP
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States